CLINICAL TRIAL: NCT04509284
Title: Effect of Resistance Training of Persistent Pain After Breast Cancer
Brief Title: Analgesic Effect of Resistance Training for Breast Cancer Survivors
Acronym: (ANTRAC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Collaborators: Danish Cancer Society (Other); Danish Cancer Survivor and Late Effects Group (Unknown); Universidad de Granada (Other)
Responsible Party: Principal Investigator, Gorm Henrik Fogh Rasmussen, Ph.D.-student, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20180090; R204-A12469 (Other Grant/Funding Number: Danish Cancer Society)
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Surgery; Chemotherapy Effect; Radiotherapy Side Effect; Pain, Chronic
Keywords: Persistent Pain; Breast cancer treatment; Physical function; Quality of life; Resistance training; Analgesic effect of resistance training of persistent pain after breast cancer (ANTRAC)
MeSH Terms: conditions — Breast Neoplasms; Radiation Injuries; Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) The statistician, who will conduct the statistical analysis, will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): Participants with persistent pain after breast cancer treatment will receive 24 sessions of individualized progressive total body resistance training, supervised by a certified strength and conditioning specialist.
  Interventions: Other: Training
- Control (Other): Participants with persistent pain after breast cancer treatment will be instructed to continue their everyday lifestyle and be encouraged not to engage in new forms of exercise or physical activity throughout the study period.
  Interventions: Other: Control

INTERVENTIONS:
Other: Training — The experimental group will perform a supervised progressive resistance training program, with five exercises for the upper- and lower body (box squat, bench press, trap bar deadlift, bench pull and lat pulldown), 2x/week for a 12 week period. The program will utilize a flexible progression system through three distinct training phases; 1) 2-4 sets of 10-12 repetitions, 2) 2-4 sets of 6-8 repetitions, 3) 2-4 sets of 2-4 repetitions. Number of sets are adjusted within session according to daily readiness while load is adjusted within and between sessions according to number of reps performed. A 3-5min rest period is provided throughout the program.
  Arms: Training
Other: Control — The control group will be instructed to continue their everyday lifestyle with no specific instruction regarding exercise and/or diet. However, they will be encouraged not to engage in new forms of exercise or physical activity throughout the study period.
  Arms: Control

SUMMARY:
Persistent pain after treatment for breast cancer is a major clinical problem, affecting 25-60 % of the patients and is a source of considerable physical disability and psychological distress. Thus, the development of novel interventions to improve pain management for these patients is of clinical importance. Resistance training (RT) is a promising tool to combat a variety of undesirable adverse effects due to breast cancer treatment. Further, research suggests that it may also be able to provide pain-relieving benefits.

Hypothesis: Resistance training will improve pain perception and physical function in the short- and long term compared to a non-training control group.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women worldwide with more than a million new cases diagnosed every year [1]. Fortunately, due to better treatment options, the population of long-term survivors is increasing. This poses new demands for knowledge on how to manage late effects to the treatment regimen. Persistent pain after treatment for breast cancer is a common and underestimated problem as well as it can be a source of considerable physical disability and psychological distress [2]. Hence, the development of novel interventions to improve pain management is of high clinical relevance. Resistance training (RT) is a promising clinical therapeutic tool to improve a variety of adverse effects to breast cancer treatment [3] and may provide several pain-relieving benefits [4]. However, the efficacy of this modality for managing persistent pain after breast cancer treatment is currently unclear. Therefore, the purpose of this project is to investigate if individualized RT can modulate persistent pain after breast cancer treatment, thereby improving our understanding of how this modality may benefit patients and contribute to clinical guidelines for pain management in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of breast cancer (grades I-IIIA).
* adult women at least 18 years of age.
* having received breast cancer treatment (i.e. surgery and possible adjuvant chemo and/or radiotherapy) at least 18 months before the start of the study.
* self reported pain in the areas of the breast, shoulder, axilla, arm and/or side of body with an intensity of ≥ 3 on a numeric rating scale (0 = no pain, 10 = worst pain imaginable).
* no signs of cancer recurrence.
* reading, writing and speaking Danish.

Exclusion Criteria:

* breast surgery for cosmetic reasons or prophylactic mastectomy.
* bilateral breast cancer.
* lymphedema.
* other chronic pain conditions (e.g., rheumatoid arthritis).
* previous diagnosis of fibromyalgia syndrome.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Change in pain sensitivity, assessed through pressure pain thresholds. | Baseline and at 3, and 6 months
  Between group comparisons of treatment effect (change in pressure pain thresholds) from baseline to follow-up) will be performed. Pressure pain thresholds will be collected with a pressure algometer with a progressive increment in pressure of 30kPa.
Change in pain intensity, assessed through a 11 point numeric rating scale (0 = no pain, 10 = worst pain imaginable). | Baseline and at 3, and 6 months
  Pain intensity is collected in two different contexts; 1) recollection for the past 3 months and 2) movement evoked pain during testing and training.

SECONDARY OUTCOMES:
Muscular strength assesses through a 1 repetition maximum (1RM) | Baseline and at 3, and 6 months
  1RM box squat, bench press, trapbar deadlift, bench pull and lat pulldown conducted in accordance with the recommendations of the American College of Sports Medicine (ACSM)
Active shoulder range of motion assessed with a universal goniometer. | Baseline and at 3, and 6 months
  Active range of motion for the affected shoulder is collected for shoulder flexion, horizontal shoulder flexion/extension, shoulder abduction and internal/external shoulder/rotation
Body composition assessed through bioelectrical impedance measurements. | Baseline and at 3, and 6 months
  Estimates of body fat mass, fat free mass, skeletal muscle mass and bodyfat percentage are collected from bioelectrical impedance using an InBody370 device.
Arm circumference measured bilaterally at a single point 30cm above the styloid process. | Baseline and at 3, and 6 months
  Arm circumference is collected to assess potential lymphedema development. A difference in circumference of >10% between arms is considered indicative of lymphedema.
Physical activity level assessed through the international physical activity questionnaire (IPAQ). | Baseline and at 3, and 6 months
  IPAQ estimates physical activity level as "low", "moderate" or "high" from the number of days and time per day conducting either hard, moderate or easy physical activity for the pas seven days.
Health related quality of life assessed through the European Organisation for Research and Treatment of Cancer (EORCT)-C30 quality of life questionaire | Baseline and at 3, and 6 months
  The EORCT-C30 QLQ estimates quality of life through a series of questions regarding the extent to which the respondee experience various restrictions in physical function and well-being common in cancer patients, ranging from 1 (not at all) to 4 (A lot) on a four point likert scale.
Quality of life assessed through the breast cancer specific European Organisation for Research and Treatment of Cancer (EORCT)-BR23 quality of life questionaire | Baseline and at 3, and 6 months
  The EORCT-C30 QLQ estimates quality of life through a series of questions regarding the extent to which the respondee experience various restrictions in physical function and well-being common in breast cancer patients, ranging from 1 (not at all) to 4 (A lot) on a four point likert scale.
Cancer fatigue assessed through the Functional Assessment of Chronic Illness Therapy (FACIT) - fatigue scale. | Baseline and at 3, and 6 months
  The FACIT-scale estimates fatigue through a series of questions regarding the extent to which the respondee experience various symptoms of fatigue, ranging from 0 (not at all) to 4 (A lot) on a five point likert scale.
Mental health assessed through the Major Depression Index (MDI) | Baseline and at 3, and 6 months
  The MDI estimates mental health through a series of questions regarding the extent to which the respondee experience various symptoms of depression, ranging from 0 (never) to 5 (All the time) on a five point likert scale.

OTHER OUTCOMES:
Summative process evaluation | At 3 months
  The summative process evaluation include the following: 1) Context of the intervention described qualitatively, 2) the dose delivered as %'age of the planed sessions effectively implemented, 3) dose received as %'age of planned sessions effectively received, 4) fidelity measured through the following items: (1) whether the training groups (i.e. same participants every session) during training sessions were consistent; (2) whether the instructors delivered all their sessions as initially scheduled; (3) whether warm-up and training were offered in accordance with the time schedules initially planned; (4) whether the time schedule were respected by participants and instructors and 5) satisfaction, rated as level of agreement with a series of statements on a five-point likert scale 1=strongly disagree, 2=disagree, 3=uncertain, 4=agree, and 5=strongly agree.
Training log, collecting daily readiness for exertion, performance, perceived exertion level and movement evoked pain. | Every session for 12 weeks.
  Daily readiness for exertion is assessed at two levels (mental and physical) prior to the warm up and each exercise on a 0-11 numeric rating scale (0 = no readiness, 10 = maximum readiness. Performance i collected as setsXrepsXload per exercise per session. Perceived level of exertion is assessed through a resistance training specific Rating of Perceived Exertion (RPE) scale based on repetitions in reserve. Movement-evoked pain is assessed per set for each exercise on a 11 point numeric rating scale (0= no pain, 10 = maximum pain).

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Madeleine, Dr. Scient, Study Chair — Aalborg University; Michael Voigt, Ph. D., Study Chair — Aalborg University; Mathias Kristiansen, Ph. D., Study Chair — Aalborg University; Manuel Arroyo-Morales, Dr. Med, Study Chair — Universidad de Granada
Locations (1):
- Department of Health Science and Technology, Aalborg University, Aalborg, Northern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cronin-Fenton DP, Norgaard M, Jacobsen J, Garne JP, Ewertz M, Lash TL, Sorensen HT. Comorbidity and survival of Danish breast cancer patients from 1995 to 2005. Br J Cancer. 2007 May 7;96(9):1462-8. doi: 10.1038/sj.bjc.6603717. Epub 2007 Apr 3. PMID 17406360
- [Background] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Background] De Backer IC, Schep G, Backx FJ, Vreugdenhil G, Kuipers H. Resistance training in cancer survivors: a systematic review. Int J Sports Med. 2009 Oct;30(10):703-12. doi: 10.1055/s-0029-1225330. Epub 2009 Jul 7. PMID 19585401
- [Background] Rice D, Nijs J, Kosek E, Wideman T, Hasenbring MI, Koltyn K, Graven-Nielsen T, Polli A. Exercise-Induced Hypoalgesia in Pain-Free and Chronic Pain Populations: State of the Art and Future Directions. J Pain. 2019 Nov;20(11):1249-1266. doi: 10.1016/j.jpain.2019.03.005. Epub 2019 Mar 21. PMID 30904519
- [Derived] Rasmussen GHF, Madeleine P, Arroyo-Morales M, Voigt M, Kristiansen M. Resistance Training-Induced Acute Hypoalgesia in Women With Persistent Pain After Breast Cancer Treatment. J Strength Cond Res. 2023 Mar 1;37(3):e16-e24. doi: 10.1519/JSC.0000000000004320. Epub 2022 Sep 28. PMID 36173261
- [Derived] Rasmussen GHF, Kristiansen M, Arroyo-Morales M, Voigt M, Madeleine P. The Analgesic Effect of Resistance Training after Breast Cancer (ANTRAC): A Randomized Controlled Trial. Med Sci Sports Exerc. 2023 Feb 1;55(2):167-176. doi: 10.1249/MSS.0000000000003034. Epub 2022 Sep 7. PMID 36084228